CLINICAL TRIAL: NCT01415661
Title: Efficacy of Cricoid Pressure in Occluding the Esophageal Entrance: A Glidescope ® Study
Acronym: CP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Procare Riaya Hospital (Other)
Responsible Party: Principal Investigator, Ahed ZEIDAN, MD, Procare Riaya Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PRH 01
Record Dates: First submitted 2011-08-04; First posted 2011-08-12 (Estimated); Last update posted 2012-04-10 (Estimated); Status verified 2012-04

CONDITIONS: Aspiration

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- obese patient (Experimental)
  Interventions: Other: cricoid pressure
- non obese patient (Experimental)
  Interventions: Other: cricoid pressure

INTERVENTIONS:
Other: cricoid pressure — The current study test by direct visual evidence the occlusion of esophageal entrance during application CP. The closure of the lumen was further demonstrated by the inability to introduce a GT into the esophagus during CP.
  Other Names: Glidescope

SUMMARY:
This investigation was designed to assess the patency of the esophageal entrance during cricoid pressure (CP) in anesthetized, paralyzed obese and non obese patients using the Glidescope ® video laryngoscope (GVL).

DETAILED DESCRIPTION:
Eighty-nine patients undergoing surgeries necessitating general anesthesia and tracheal intubation were enrolled in this study. Group 1 (OB) including obese patients (n= 59) was undergoing bariatric surgery. Following rapid sequence induction/intubation (RSII) anesthesia with cricoid pressure, clear view of the vocals cord and the entrance to the esophagus were assessed using Glidescope® video laryngoscope before intubation and following intubation. Following securing the airway, efficacy of cricoid pressure was tested by the capability to insert gastric tubes (20 and 38 Fr) under direct vision using GVL. Group 2 (NOB) including non-obese patients (n=30) was undergoing moderate surgery requiring tracheal intubation under general anesthesia. Efficacy of cricoid pressure was also tested similarly using GT's (20 and 38 Fr) following induction of anesthesia and before intubation. Inability of GT insertion was recorded as non-patent esophagus (effective CP) and successful insertion of GT was recorded as patent esophagus (ineffective CP). Then CP was released and insertion of GT achieved for correct verification of the esophageal opening position in both groups.

ELIGIBILITY:
Inclusion Criteria:

* Obese patients ( BMI 40-70 kg/m2)
* No Contre indication to cricoid pressure
* No-obese patients (BMI < 40)

Exclusion Criteria:

* ASA 3 and 4
* Contre indication to cricoid pressure

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 89 (Actual)
Dates: Start 2011-01; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Efficacy of Cricoid Pressure for Prevention of Aspiration | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: AHED ZEIDAN, MD, Study Chair — Procare Riaya Hospital
Locations (1):
- procare Riaya Hospital, Khobar, Estern, Saudi Arabia